CLINICAL TRIAL: NCT03202082
Title: Impact of Neuropsychological Evaluation on Epilepsy Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Satisfaction after Evaluation
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuropsychological testing (Experimental): Participants from this group will be administered a neuropsychological battery in addition to the initial and follow-up surveys
  Interventions: Behavioral: Neuropsychological testing
- Treatment as usual (No Intervention): Participants from this group will be administered the initial and follow-up survey.

INTERVENTIONS:
Behavioral: Neuropsychological testing — Neuropsychological testing evaluates various aspects of a participants cognitive ability as well as mood.
  Arms: Neuropsychological testing

SUMMARY:
The present study aims to expand the evidence base of neuropsychological services in the context of medical management of epilepsy, examining whether treatment outcome and patient satisfaction with medical care are significantly improved when neuropsychological evaluation is included as an additional component of medical care within a comprehensive epilepsy center. All participants will complete an initial survey and a follow-up survey regarding views towards their epilepsy treatment. Participants will be randomized into one of two groups. One group will be given a neuropsychological battery in addition to the survey. The primary study hypothesis is that the addition of neuropsychological services to treatment-as-usual will result in significant improvements in (a) satisfaction with medical care, (b) patient perceived treatment outcome, and (c) physician-rated medical compliance. The secondary hypothesis is that participants who undergo neuropsychological evaluation will be generally satisfied with their experience with neuropsychological services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* experiencing some degree of epilepsy-related symptoms, but not of such severity as to preclude them from being able to provide consent or undergo neuropsychological assessment (requiring extended inpatient treatment, severely aphasic, or MMSE score < 25)

Exclusion Criteria:

* Previously undergone neuropsychological testing
* Currently pursuing surgical treatment for epilepsy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Epilepsy Outcome Study Survey | 2-4 months
  A brief questionnaire regarding the participants views on their epilepsy treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No